CLINICAL TRIAL: NCT06847217
Title: Effect of Applying Oral Hygiene Care on Swallowing in Stroke Patients With Oropharyngeal Dysphagia: A Multi-Arm Randomized Controlled Trial
Brief Title: Effect of Applying Oral Hygiene Care on Swallowing in Stroke Patients With Oropharyngeal Dysphagia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ONZ-2024-0245
Record Dates: First submitted 2025-02-05; First posted 2025-02-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Dysphagia After Stroke
Keywords: Stroke; Deglutition; Dysphagia; Oral care; Swallowing disorder
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: This study was designed as a multi-arm randomized controlled trial (RCT) comprising four groups: a control group, a mouth moisturization group, a mechanical oral hygiene group, and a combined care group. Patients in each group will be blinded to the intervention, and the primary outcomes measured by the test of masticating and swallowing solids (TOMASS) will be recorded and sent to a blinded examiner.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Patients will receive oral cleaning using only water and gauze as a usual process.
- Mouth moisturization group (Experimental): Patients will undergo oral cleaning with a water-based hydrating gel.
  Interventions: Other: Mouth moisturization
- Mechanical oral hygiene group (Experimental): Patients with natural teeth/or denture will receive oral care using a mechanical oral hygiene care.
  Interventions: Other: Mechanical oral hygiene care
- Combined care group (Experimental): Patients will receive a comprehensive oral hygiene intervention incorporating mouth cleaning, mechanical oral hygiene, and moisturization.
  Interventions: Other: Combined care

INTERVENTIONS:
Other: Mouth moisturization — This intervention will include mouth cleaning with water and gauze to remove plaque and debris. Water-based hydrating gels (bioXtra Dry Mouth Oral Gel, Lifestream Pharma N.V., Seneffe, Belgium) will be then applied to all oral structures, including the lips, tongue, palate, and cheeks, using gloved fingers or a small toothbrush. In the presence of dried secretions, the gels will be massaged into these areas and left to act for a few minutes to facilitate removal and reduce patient discomfort.
  Arms: Mouth moisturization group
Other: Mechanical oral hygiene care — Patients with natural teeth will be treated using a soft toothbrush and a sodium lauryl sulfate-free fluoride toothpaste (meridol® toothpaste, Colgate-Palmolive Company, Belgium). The teeth will be brushed using the modified BASS technique. Subsequently, the tongue will be cleaned with either a scraper. For participants wearing dentures, the dentures will be cleaned using a denture brush and soap.
  Arms: Mechanical oral hygiene group
Other: Combined care — Patients will receive a comprehensive oral hygiene intervention incorporating mouth cleaning, mechanical oral hygiene, and moisturization. The procedure will begin with oral cleaning using water and gauze, followed by mechanical oral hygiene, and conclude with the application of the hydrating gel.
  Arms: Combined care group

SUMMARY:
Post-stroke dysphagia (PSD) is a common condition, affecting over 40% of patients within hours to days following a stroke. It is associated with negative outcomes, including higher rates of mortality and dependency, incidence of aspiration, pneumonia, and malnutrition. The presence of dysphagia, combined with poor oral health, significantly increases the risk of these adverse outcomes. However, there is limited knowledge regarding the impact of oral care practices on these outcomes, as well as their effect on oral function and swallowing in acute stroke patients.

The optimal approach to delivering oral care remains undefined, and practices vary widely among healthcare professionals. Many providers often avoid using toothbrushes or toothpaste due to concerns about the risk of aspiration, despite recommendations for their use. Electric and suction toothbrushes may offer effective alternatives, but their high cost and uncertain benefits in the context of an acute stroke pose challenges.

This study aims to measure the immediate effects of three different oral hygiene protocols: on masticatory and swallowing abilities in stroke patients with oropharyngeal dysphagia during the acute and subacute phases. The protocols are mouth moisturization, mechanical oral hygiene, and combined care (mouth moisturization and mechanical oral hygiene). The primary objective is to evaluate the effect of combined care compared to a control group with care as usual. The secondary objective is to evaluate the other 2 oral hygiene protocols relative to combined care.

DETAILED DESCRIPTION:
Data collection:

1. At trial baseline (Before oral hygiene intervention)

   * 1.1. Socio-demographic data: age, gender, education, living conditions, and allowance for increased health care cost reimbursement
   * 1.2. Medical information: smoking habit, medications, and medical background such as stroke type and location, stroke history, National Institutes of Health Stroke Scale (NIHSS), and Functional Oral Intake Scale (FOIS),
   * 1.3. Dental information from oral examination:
   * Oral care ability
   * Oral hygiene index including dental plaque, tongue plaque, and denture plaque.
   * Oral disease: Periodontal status and sign of periodontitis as tooth mobility, clinical dental caries, and clinical mucosal lesions.
   * Oral status: the number of functional teeth, the number of posterior occluding pairs, and denture status
   * Clinical oral dryness scoring
   * 1.4. Tongue strength using maximum isometric pressure (MIP) from the Iowa Oral Performance Instrument (IOPI) during rest and swallowing stages
   * 1.5. Test of Masticating and Swallowing Solids (TOMASS): number of discrete bites, number of masticatory cycles, number of swallows, and total time
   * 1.6. Oral residue score (ORS)
2. After oral hygiene intervention

   * 2.1. Clinical measurements
   * Modified TOMASS by using a half cracker: number of discrete bites, number of masticatory cycles, number of swallows, and total time
   * Tongue strength using MIP from IOPI during rest and swallowing stages
   * ORS
   * 2.2. Subjective measurements: Visual Analogue Scale (VAS)

Sample size:

Sample size calculations were based on both the primary and secondary objectives, focusing on the primary outcomes: number of masticatory cycles, number of swallows, and total time.

For both objectives, sample size estimation was conducted using an independent t-test to compare means in a superiority test between two groups, with an alpha level of 0.05 and a power of 0.80. G*Power software (version 3.1.9.2, Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany) was used for the calculation. The effect size for the intervention was estimated based on the standard deviation (SD) from pilot data, combined with the clinically relevant mean difference determined by the research team using pilot data and previous studies comparing individuals with dysphagia to healthy individuals.

The required sample size, calculated using the smallest effect size corresponding to total time in the primary and secondary objectives, was 53 and 62 participants per group, respectively. These calculations were based on an SD of 40.2 with a clinically relevant mean difference of 22 seconds for the primary objective, and an SD of 21.7 with a clinically relevant mean difference of 11 seconds for the secondary objective.

To account for a 5% dropout rate, the final sample size was adjusted to 65 participants per group, resulting in a total of 260 participants.

Randomization:

Randomization was conducted using a 1:1:1:1 allocation ratio with variable block sizes of 4 and 8, with sequences independently generated using Microsoft Excel version 16 (Microsoft, New Mexico, USA). Allocation and data collection were managed through REDCap (Research Electronic Data Capture), hosted at Ghent University Hospital.

Statistical methods:

The primary analysis will evaluate the superiority of the combined care group over the control group. If statistical significance is achieved, a secondary analysis will compare the combined care group with the mechanical oral hygiene and mouth moisturization groups, respectively.

An exploratory analysis using hierarchical pairwise comparisons will be conducted if both comparisons in the secondary analysis and the statistical analysis across all four groups show significance. The pairwise comparisons will be ordered sequentially, first comparing the mouth moisturization group with the control group, then the mechanical oral hygiene group with the control group and finally comparing the mouth moisturization and mechanical oral hygiene groups with each other.

All analyses will be performed using analysis of covariance (ANCOVA), with pre-intervention outcomes as covariates and a significance level of 0.05.

To address missing data, multiple imputation will be applied. Sensitivity analyses will compare results from imputed data with those from complete case analysis to ensure the robustness of findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the stroke unit at Ghent University and diagnosed with oropharyngeal dysphagia.
* Agreement to participate in the study and having signed an informed consent form.
* Age over 18 years.
* Sufficient cognitive abilities and language skills to understand the swallowing exercises.

Exclusion Criteria:

* A history of surgical intervention on the tongue.
* Edentulous individuals, both fully edentulous or edentulous in one dental arch, if they do not wear dentures.
* Patients with a penetration-aspiration scale (PAS) of 7 or 8 under flexible endoscopic evaluation of swallowing (FEES), at the international dysphagia diet standardisation initiative (IDDSI) level 7.
* Patients who cannot perform TOMASS, indicated by 25% or more of the amount of cracker's bolus that can be considered as the same cracker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Test of Mastication and Swallowing Solids (TOMASS): number of masticatory cycles | Before the intervention (baseline period) and immediately after the intervention on the same day.
  This outcome assesses mastication and swallowing efficiency by counting the number of masticatory cycles, using half the standard amount of a cracker.
Test of Mastication and Swallowing Solids (TOMASS): number of swallows | Before the intervention (baseline period) and immediately after the intervention on the same day.
  This outcome assesses mastication and swallowing efficiency by counting the number of swallows, using half the standard amount of a cracker.
Test of Mastication and Swallowing Solids (TOMASS): total time | Before the intervention (baseline period) and immediately after the intervention on the same day.
  This outcome assesses mastication and swallowing efficiency by recording the total time (seconds) taken to consume half the standard amount of a cracker.

SECONDARY OUTCOMES:
Test of Mastication and Swallowing Solids (TOMASS): number of discrete bites | Before the intervention (baseline period) and immediately after the intervention on the same day.
  This outcome assesses mastication and swallowing efficiency by counting the number of discrete bites, using half the standard amount of a cracker.
Tongue strengthening performance | Before the intervention (baseline period) and immediately after the intervention on the same day.
  This outcome assesses patients' ability to generate anterior maximum isometric pressure (MIP) during both the resting and swallowing stages, using the Iowa Oral Performance Instrument (IOPI).
Oral residue score (ORS) | Before the intervention (baseline period) and immediately after the intervention on the same day.
  The outcome assesses the oral residue remaining in patients' mouth after the TOMASS method, using a 4-point scale (0-3) to evaluate oral residue after eating a cracker in eight areas of the mouth, including the left teeth, right teeth, left sulcus and cheek, right sulcus and cheek, hard palate, soft palate, dorsum of the tongue, and floor of the mouth with a total score of 24.
Patient's subjective measurements | Before the intervention (baseline period) and immediately after the intervention on the same day.
  This outcome assesses the patient's experience in 9 topics using the Visual Analogue Scale (VAS), a 0-100 mm scale, where the 0-100 score indicates the patient's experience. The highest score could represent either worse or better experiences depending on each topic. The assessed topics include:
  * I cough when I eat a cracker
  * Chewing a cracker is easy
  * Swallowing a cracker is difficult
  * I experience pain when swallowing a cracker
  * There is food left in my mouth after eating a cracker
  * Placing the bulb in the correct location in my mouth is easy (for IOPI)
  * Pushing the bulb is difficult (for IOPI)
  * My mouth is dry
  * I have a pleasant feeling in my mouth

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Janssens, Principal Investigator — Ghent University, Ghent, Belgium
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
The IPD must be shared as anonymized or pseudonymized information, which may be included in a meta-analysis upon request. Data transfer must be conducted under Ghent University Hospital conditions, with legal experts drafting and reviewing the agreement (https://hiruz.be/cu/). Additionally, any data containing personal information requires approval from the Ethics Committee before transfer.

REFERENCES:
- [Background] Das P, Challacombe SJ. Dry Mouth and Clinical Oral Dryness Scoring Systems. Prim Dent J. 2016 Feb 1;5(1):77-79. doi: 10.1177/205016841600500110. PMID 29029657
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Wu CP, Tu YK, Lu SL, Chang JH, Lu HK. Quantitative analysis of Miller mobility index for the diagnosis of moderate to severe periodontitis - A cross-sectional study. J Dent Sci. 2018 Mar;13(1):43-47. doi: 10.1016/j.jds.2017.11.001. Epub 2018 Feb 3. PMID 30895093
- [Background] Van der Velden U. The Dutch periodontal screening index validation and its application in The Netherlands. J Clin Periodontol. 2009 Dec;36(12):1018-24. doi: 10.1111/j.1600-051X.2009.01495.x. PMID 19929955
- [Background] Janssens LE, Temmerman E, Maertens J, De Visschere L, Petrovic M, Janssens BE. A comparative analysis of oral hygiene in nursing homes with and without a structured oral healthcare programme. Gerodontology. 2025 Mar;42(1):78-85. doi: 10.1111/ger.12773. Epub 2024 Jun 21. PMID 39959995
- [Background] Franciotti R, Di Maria E, D'Attilio M, Aprile G, Cosentino FG, Perrotti V. Quantitative Measurement of Swallowing Performance Using Iowa Oral Performance Instrument: A Systematic Review and Meta-Analysis. Biomedicines. 2022 Sep 18;10(9):2319. doi: 10.3390/biomedicines10092319. PMID 36140420
- [Background] Todaro F, Pizzorni N, Scarponi L, Ronzoni C, Huckabee ML, Schindler A. The Test of Masticating and Swallowing Solids (TOMASS): Reliability and validity in patients with dysphagia. Int J Lang Commun Disord. 2021 May;56(3):558-566. doi: 10.1111/1460-6984.12613. Epub 2021 Mar 9. PMID 33687133
- [Background] Huckabee ML, McIntosh T, Fuller L, Curry M, Thomas P, Walshe M, McCague E, Battel I, Nogueira D, Frank U, van den Engel-Hoek L, Sella-Weiss O. The Test of Masticating and Swallowing Solids (TOMASS): reliability, validity and international normative data. Int J Lang Commun Disord. 2018 Jan;53(1):144-156. doi: 10.1111/1460-6984.12332. Epub 2017 Jul 5. PMID 28677236
- [Background] Cohen DL, Roffe C, Beavan J, Blackett B, Fairfield CA, Hamdy S, Havard D, McFarlane M, McLauglin C, Randall M, Robson K, Scutt P, Smith C, Smithard D, Sprigg N, Warusevitane A, Watkins C, Woodhouse L, Bath PM. Post-stroke dysphagia: A review and design considerations for future trials. Int J Stroke. 2016 Jun;11(4):399-411. doi: 10.1177/1747493016639057. Epub 2016 Mar 22. PMID 27006423